CLINICAL TRIAL: NCT03671096
Title: A Prospective Multi Center Clinical Study to Evaluate the Safety And Effectiveness of the Transform™ Corneal Allograft (TCA) for Treatment of Hyperopia
Brief Title: Safety and Efficacy of the Transform™ Corneal Allograft for Hyperopia Correction
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: The sponsor determined at one study (PRO-010) was sufficient
Sponsor: Allotex, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PRO_012
Record Dates: First submitted 2018-09-06; First posted 2018-09-14 (Actual); Last update posted 2020-03-11 (Actual); Status verified 2020-03

CONDITIONS: Hyperopia
Keywords: Intrastromal; Corneal; Allograft
MeSH Terms: conditions — Hyperopia

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intrastromal TCA Inlay (Experimental): Implant Intrastromal TCA using femto-second laser surgery It is expected to be carried out once only during the study duration
  Interventions: Other: Intrastromal TCA Inlay

INTERVENTIONS:
Other: Intrastromal TCA Inlay — An intrastromal inlay that will be provided to correct the required hyperopic correction

SUMMARY:
The objective of this clinical study is to evaluate the safety and effectiveness of intrastromal implantation of the Allotex TCA for improving distance vision in hyperopic subjects.

The overall objective with respect to visual outcome is to provide improved vision without the requirement of additional visual aids.

DETAILED DESCRIPTION:
This research provides a method to primarily correct refractive error by implanting a natural tissue graft. The level of correction will range from +1.00 to +6.00D which represents a range of refractive error that is difficult to manage using the same refractive surgical techniques used to correct myopia.

The other objective is to assess graft tolerance and safety so it can be applied to subjects that require other forms of visual correction.

This technique also permits the potential for graft removal if required and the patient should revert back to their previous prescription as no tissue is removed when applying this technique.

Beginning in 1949 with the pioneering work of Jose Barraquer, there has been an interest in using natural corneal tissue to change the refractive properties of the eye. In recent years, non-allogenic, synthetic corneal implants have received marketing approval in the United Stated and Europe for refractive purposes. Although synthetic implants are made of biocompatible materials they are not equivalent to an allogenic implant in terms of biocompatibility. The Allotex TCA is a piece of acellular cornea, sterilized with electron beam radiation and shaped to a particular shape using a laser. The availability of precise laser shaping systems and sterile corneas are the key factors that make the use of allogenic implants possible.

The implant is placed on the posterior surface of Bowmans layer of the cornea, in a corneal flap formed by a femtosecond laser.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must have signed the written informed consent form and been given a copy.
* 21 years of age or older on the day the surgery is performed.
* Best distance corrected visual acuity of 20/20 or better in both eyes.
* Near visual acuity correctable to at least 20/20 in both eyes.
* Manifest refraction spherical equivalent (MRSE) between +1.00 and +6.00 D with no more than 0.75 D of refractive cylinder in both eyes.
* Stable vision, i.e. MSRE within 0.50 D over prior 12 months in both eyes.
* Contact lens wearers must discontinue hard or rigid gas permeable lenses for at least 2 weeks and discontinue soft lenses for at least 3 days prior to baseline examination in both eyes.
* Contact lens wearers must have two (2) central keratometry readings with regular mires and two (2) manifest refractions taken at least one week apart, with no contact lens wear between. Keratometric values must not differ by more than ±0.50 D in any meridian and MRSE values must not differ more than ±0.50 D in both eyes.
* Average corneal power of ≥ 41.00 D and ≤ 47.00 D in both eyes.
* Anticipated postoperative average corneal power (preoperative average corneal power + intended correction) ≤ 50.00 D in both eyes.
* Subjects must be willing and able to return for scheduled follow-up examinations for 24 months after surgery of the fellow eye.

Exclusion Criteria:

* Difference of > 0.75 D between the manifest refraction spherical equivalent and the cycloplegic refraction spherical equivalent in either eye.
* Anterior segment pathology in either eye.
* Signs or symptoms of clinically significant cataracts in either eye.
* Residual, recurrent, active ocular or uncontrolled eyelid disease, or any corneal abnormality (including endothelial dystrophy, recurrent corneal erosion, etc.) in either eye.
* Central corneal thickness <470 microns in either eye.
* Residual stromal thickness of <300 microns in either eye.
* Topographic signs of keratoconus (or keratoconus suspect) or other ectatic disorders in either eye.
* Subjects with clinically significant dry eyes, as determined by Tear Breakup Time (TBUT) of < 7 seconds or the presence of greater than mild symptoms of dryness or discomfort or SPK greater than grade 1.
* Distorted or unclear corneal mires on topography maps of either eye.
* Macular degeneration, retinal detachment, or any other fundus pathology that would prevent an acceptable visual outcome in either eye.
* Any prior ocular surgery in either eye.
* History of herpes zoster or herpes simplex keratitis in either eye.
* History of steroid-responsive rise in intraocular pressure (IOP), preoperative IOP >21 mm Hg, glaucoma, or are a glaucoma suspect in either eye.
* Using systemic medications with significant ocular side effects.
* Pregnant, lactating, or planning to become pregnant during the course of the study.
* Known sensitivity to planned study concomitant medications.
* Participating in any ophthalmic drug or device clinical trial during the time of this clinical investigation.

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2018-10 (Estimated); Primary Completion 2021-01 (Estimated); Study Completion 2021-01 (Estimated)

PRIMARY OUTCOMES:
Assessment of the accuracy and stability of hyperopia refractive correction following intervention with the Transform™ Corneal Allograft inlay. | 6 months
  The primary effectiveness endpoint is predictability of the refractive error within ±1.00 D of the intended refractive outcome at 6 months post-operatively. A minimum of 65% of eyes should have an achieved manifest refraction within ±1.00 D of the intended refractive outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Slade, MD, Study Director — Study Medical Monitor/Consultant
Locations (11):
- Austria (2):
  - Gemini Augenlaser Wien, Vienna, Opernring 1
  - Sekhraft Augenzentrum Wien, Vienna
- Medipolis Wilrijk, Antwerp, Boomsesteenweg 223, Belgium
- France (2):
  - Hospital Pierre Paul Riquet, Toulouse, Purpan
  - Institute Laser Vision Noemie de Rothschild, Fondation Ophthalmolique Adolphe de Rothschild, Paris
- Wellington Eye Clinic, Dublin, Beacon Court Sandyford, Ireland
- Switzerland (2):
  - Laser Vista, Basel
  - Eye Clinic Orasis AG, Reinach
- United Kingdom (3):
  - Optegra Eye Hospital, London, Marylebone
  - Corneo Plastic Unit and Eye Bank Queen Victoria Hospital, East Grinstead
  - Centre for Sight, London